CLINICAL TRIAL: NCT00827073
Title: The Effects on Betadine 5% Penetration When Using Lidocaine 2% Jelly Versus Topical Tetracaine 0.5% for Topical Phacoemulsification Cataract Surgery.
Brief Title: Comparison of Tetracaine 0.5% and Lidocaine 2% Jelly for Topical Phacoemulsification Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hermann Eye Center (Other)
Responsible Party: Principal Investigator, Joseph Selem, Principle Investigator, Hermann Eye Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-MS-08-0454
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Lidocaine; Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetracaine 0.5% drop (Active Comparator): Tetracaine 0.5% drop of betadine will be used on the operative eye after Tetracaine has been administered
  Interventions: Drug: tetracaine 0.5%
- Lidocaine 2% Jelly (Active Comparator): Lidocaine 2% Jelly drop of betadine will be used on the operative eye after Lidocaine 2% Jelly has been administered
  Interventions: Drug: Lidocaine 2% Jelly

INTERVENTIONS:
Drug: tetracaine 0.5% — betadine 5%
  Arms: Tetracaine 0.5% drop
Drug: Lidocaine 2% Jelly — Betadine 5%
  Arms: Lidocaine 2% Jelly

SUMMARY:
The purpose of this study is to determine if there is a difference on the penetration of betadine 5% when using lidocaine 2% jelly versus topical tetracaine 0.5% in topical cataract surgery. This will be assessed comparing bacterial colony count and species by taking swabs from the eye surface before and after the topical anesthesia has been administered.

DETAILED DESCRIPTION:
The purpose of this research study is to show that using Lidocaine2% jelly before surgery as an anesthetic (keep you from feeling touch or pain) for cataract surgery does not block the antiseptic (cleans and kills germs) effect of Betadine5%.

ELIGIBILITY:
Inclusion Criteria:

* greater or equal to 18 years old
* uni- or bi-lateral visually significant cataracts

Exclusion Criteria:

* hypersensitivity to betadine5%, topical tetracaine0.5%, or lidocaine2% jelly
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nan Wang, MD, Principal Investigator — Robert Cizik Eye Clinic and Department of Ophthalmology and Visual Science at The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Plaza Surgery Center, Houston, Texas, United States

REFERENCES:
- [Background] Fichman RA. Use of topical anesthesia alone in cataract surgery. J Cataract Refract Surg. 1996 Jun;22(5):612-4. doi: 10.1016/s0886-3350(96)80019-8. PMID 8784636
- [Background] Roman S, Auclin F, Ullern M. Topical versus peribulbar anesthesia in cataract surgery. J Cataract Refract Surg. 1996 Oct;22(8):1121-4. doi: 10.1016/s0886-3350(96)80129-5. PMID 8915811
- [Background] Virtanen P, Huha T. Pain in scleral pocket incision cataract surgery using topical and peribulbar anesthesia. J Cataract Refract Surg. 1998 Dec;24(12):1609-13. doi: 10.1016/s0886-3350(98)80351-9. PMID 9850899
- [Background] Bellucci R. Anesthesia for cataract surgery. Curr Opin Ophthalmol. 1999 Feb;10(1):36-41. doi: 10.1097/00055735-199902000-00007. PMID 10387317
- [Background] Amiel H, Koch PS. Tetracaine hydrochloride 0.5% versus lidocaine 2% jelly as a topical anesthetic agent in cataract surgery: comparative clinical trial. J Cataract Refract Surg. 2007 Jan;33(1):98-100. doi: 10.1016/j.jcrs.2006.09.013. PMID 17189801
- [Background] Leong JK, Shah R, McCluskey PJ, Benn RA, Taylor RF. Bacterial contamination of the anterior chamber during phacoemulsification cataract surgery. J Cataract Refract Surg. 2002 May;28(5):826-33. doi: 10.1016/s0886-3350(01)01160-9. PMID 11978463
- [Background] Ciulla TA, Starr MB, Masket S. Bacterial endophthalmitis prophylaxis for cataract surgery: an evidence-based update. Ophthalmology. 2002 Jan;109(1):13-24. doi: 10.1016/s0161-6420(01)00899-5. PMID 11772573
- [Background] Speaker MG, Menikoff JA. Prophylaxis of endophthalmitis with topical povidone-iodine. Ophthalmology. 1991 Dec;98(12):1769-75. doi: 10.1016/s0161-6420(91)32052-9. PMID 1775308
- [Background] Deramo VA, Lai JC, Fastenberg DM, Udell IJ. Acute endophthalmitis in eyes treated prophylactically with gatifloxacin and moxifloxacin. Am J Ophthalmol. 2006 Nov;142(5):721-5. doi: 10.1016/j.ajo.2006.05.044. Epub 2006 Sep 20. PMID 16989762
- [Background] Maclean H, Burton T, Murray A. Patient comfort during cataract surgery with modified topical and peribulbar anesthesia. J Cataract Refract Surg. 1997 Mar;23(2):277-83. doi: 10.1016/s0886-3350(97)80354-9. PMID 9113582
- [Background] Patel BC, Clinch TE, Burns TA, Shomaker ST, Jessen R, Crandall AS. Prospective evaluation of topical versus retrobulbar anesthesia: a converting surgeon's experience. J Cataract Refract Surg. 1998 Jun;24(6):853-60. doi: 10.1016/s0886-3350(98)80143-0. PMID 9642600
- [Background] Seal DV, Barry P, Gettinby G, Lees F, Peterson M, Revie CW, Wilhelmus KR; ESCRS Endophthalmitis Study Group. ESCRS study of prophylaxis of postoperative endophthalmitis after cataract surgery: Case for a European multicenter study. J Cataract Refract Surg. 2006 Mar;32(3):396-406. doi: 10.1016/j.jcrs.2006.02.014. PMID 16631046
- [Background] Ferguson AW, Scott JA, McGavigan J, Elton RA, McLean J, Schmidt U, Kelkar R, Dhillon B. Comparison of 5% povidone-iodine solution against 1% povidone-iodine solution in preoperative cataract surgery antisepsis: a prospective randomised double blind study. Br J Ophthalmol. 2003 Feb;87(2):163-7. doi: 10.1136/bjo.87.2.163. PMID 12543744

RESULTS

PARTICIPANT FLOW:
Groups:
- Tetracaine 5% Drop: betadine: betadine 5%, topical anesthetic drop
- Lidocaine 2% Jelly: betadine: betadine 5% Anesthetic: lidocaine 2% jelly
Period: Overall Study
Arm/Group | Tetracaine 5% Drop | Lidocaine 2% Jelly
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tetracaine 5% Drop: betadine: betadine 5%
  topical anesthetic
- Lidocaine 2% Jelly: betadine: betadine 5%
  anesthetic
- Total: Total of all reporting groups
Arm/Group | Tetracaine 5% Drop | Lidocaine 2% Jelly | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: year] | 70.0 (7.4) | 68.4 (11.8) | 69.2 (9.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 14 | 12 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Ln(Bacterial Colony Count) From Pre-antibiotic Administration to Post Study Medication Swabs
Description: Within 3 hours from time of culture acquisition, the samples will be vortexed for 30 seconds and 100µl aliquots will be plated onto 5% sheep blood and chocolate agar plates. These plates will be incubated with 5% carbon dioxide at 35˚ C for 72 hours. After 72 hours all plates will be read for colony count and identification of all isolates will be performed using routine microbiological methods. The natural log of bacterial bacterial colony count will be used for the outcome measure.
Time Frame: (1) Pre-antibiotics swab, and (2) Post-study medication (pre surgery)
Measure: Mean (Standard Deviation); unit: Ln(bacterial colony count)
Groups:
- Tetracaine 0.5% Drop: betadine: betadine 5%
  topical anesthetic
Arm/Group | Tetracaine 0.5% Drop | Lidocaine 2% Jelly
Number analyzed (Participants) | 20 | 20
Ln(bacterial colony count) | -0.14 (0.67) | -0.52 (1.85)

2. Primary Outcome: Number of Bacterial Species in Pre-antibiotic Administration and in Post Study Medication Swabs
Time Frame: (1) Pre-antibiotics swab and (2) Post-study medication (pre surgery)
Measure: Mean (Standard Deviation); unit: bacterial spceies
Arm/Group | Tetracaine 0.5% Drop | Lidocaine 2% Jelly
Number analyzed (Participants) | 20 | 20
bacterial spceies
  pre number of bacterial spices | 1 (0) | 1 (0)
  post surgery number of bacterial speices | 1 (0) | 1 (0)

ADVERSE EVENTS:
Arm/Group | Tetracaine 0.5% Drop | Lidocaine 2% Jelly
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No